CLINICAL TRIAL: NCT06737354
Title: An Exploratory Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of IVB103 Injection in Subjects With Neovascular (Wet) Agerelated Macular Degeneration (nAMD).
Brief Title: Safety and Efficacy Study of IVB103 Injection in Subjects With Neovascular (Wet) Agerelated Macular Degeneration (nAMD).
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: InnoVec Biotherapeutics Inc. (Industry)
Collaborators: NeoVec Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IVB103-C101
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: nAMD
Keywords: nAMD; Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- IVB103 Treatment Arm（Low dose） (Experimental): Intraocular injection of a single low dose of IVB103
  Interventions: Genetic: IVB103 Injection（Low dose）
- IVB103 Treatment Arm（Intermediate dose） (Experimental): Intraocular injection of a single intermediate dose of IVB103
  Interventions: Genetic: IVB103 Injection（Intermediate dose）
- IVB103 Treatment Arm（High dose） (Experimental): Intraocular injection of a single high dose of IVB103
  Interventions: Genetic: IVB103 Injection（High dose）

INTERVENTIONS:
Genetic: IVB103 Injection（Low dose） — Single intravitreal injection
  Arms: IVB103 Treatment Arm（Low dose）
Genetic: IVB103 Injection（Intermediate dose） — Single intravitreal injection
  Arms: IVB103 Treatment Arm（Intermediate dose）
Genetic: IVB103 Injection（High dose） — Single intravitreal injection
  Arms: IVB103 Treatment Arm（High dose）

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of IVB103 injection in subjects with nAMD.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center dose escalation study. One eye of each participant will receive a single IVB103 injection by intravitreal injection. Participants will be followed for 52 weeks after which they will continue to be followed for up to 5 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate and sign the informed consent form;
2. Age≥ 50 years old, gender is not limited;
3. Confirmed presence of active CNV secondary to nAMD in the macula of study eye;
4. The total area of all types of lesions in the study eye < 30 mm2;
5. The Best Corrected Visual Acuity (BCVA) detected by the Early Treatment Diabetic Retinopathy Study (ETDRS) eye chart in the study eye is 63~19 letters (including boundary values), which is equivalent to 20/63 to 20/400 of the Snellen Eye Chart;
6. The BCVA detected by the ETDRS eye chart in the non-study eye is not less than 19 letters, which is equivalent to 20/400 of the Snellen Eye Chart;
7. The study eye has received at least 2 episodes of intravitreal anti- VEGF therapy within 6 months prior to screening and has responded within two weeks of the lead-in period of anti-VEGF standard therapy (Aflibercept injection);
8. At screening, the blood pregnancy test result of females of childbearing potential (e.g., females who have not undergone surgical sterilization or less than 1 year after menopause) is negative. Male and female subjects of childbearing potential agree to use effective contraception throughout the study and for at least 12 months after dosing.

Exclusion Criteria:

Study Eye：

1. Opacity of refractive media or inability to dilate pupils in the study eye that significantly interferes with visual acuity detection, anterior segment or fundus assessment;
2. Presence of retinal hemorrhage, geographic atrophy, scarring or fibrosis, dense subfoveal hard exudate, retinal pigment epithelium (RPE) tear involving the fovea in the study eye;
3. The study eye is combined with ocular diseases that affect central vision (e.g., diabetic retinopathy, retinal vein occlusion, vascular streaks, pathological myopia, retinal detachment, macular hole, epimacular membrane, toxoplasmosis, optic nerve disease, central serous choroidopathy, Inherited Retinal Diseases(IRDs), etc.);
4. Active intraocular or periocular infection (such as blepharitis, conjunctivitis, keratitis, scleritis, etc.) in the study eye;
5. Patients with glaucoma and ocular hypertension (intraocular pressure ≥ 25mmHg during the screening period) in the study eye;
6. Subjects with a history of intravitreal procedures other than anti- VEGF administration within the last six months (e.g., vitrectomy, macular translocation, trabecular meshwork removal, or other filtration surgery;
7. History of laser or photodynamic therapy for nAMD;
8. Presence of an ocular implant in the study eye (excluding intraocular lens, custom flex iris prosthesis); Either eye：
9. History of uveitis in either eye; Systemic diseases and others：
10. Those with diffuse intravascular coagulation and obvious bleeding tendency (such as hemoptysis, hematemesis, severe purpura, etc.) within 3 months before screening;
11. History of myocardial infarction, unstable angina, coronary revascularization, cerebrovascular accident (including TIA), history of other thromboembolic diseases (such as thromboembolic angiitis, pulmonary embolism, deep vein thrombosis, portal vein thrombosis, etc.), New York Heart Association (NYHA) grade ≥ II cardiac insufficiency, severe unstable ventricular arrhythmia, within 6 months prior to screening;
12. Have contraindications to transient immunosuppression of systemic prophylaxis (including but not limited to tuberculosis, osteoporosis, peptic ulcer, severe affective disorder) or immunocompromised;
13. Patients with systemic immune diseases (including systemic lupus erythematosus, ankylosing spondylitis, rheumatoid arthritis, etc.);
14. Diabetic patients with any of the following conditions: Known macrovascular complications; Glycosylated hemoglobin at screening（HbA1c）>7.5%; Those who have received more than two oral hypoglycemic drugs or received insulin or GLP-1 receptor agonists therapies;
15. Hypertensive patients with poor blood pressure control (defined as:

    systolic blood pressure ≥ 160 mmHg or diastolic blood pressure

    ≥100 mmHg when the subject is seated after receiving antihypertensive medication);
16. Any uncontrollable clinical illness (such as severe psychiatric, respiratory and other systemic diseases and history of malignant tumors);
17. Patients with abnormal liver and kidney function: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal; Total bilirubin ≥ 1.5 times the upper limit of normal, creatinine and urea/urea nitrogen ≥ 1.5 times the upper limit of normal;
18. Patients with abnormal coagulation function: prothrombin time (PT) > upper limit of normal value of 3 seconds or activated partial thromboplasting time (APTT) > upper limit of normal value of 10 seconds; Haemoglobin (HGb) < 10 g/dL;
19. Those who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, treponema pallidum antibody and human immunodeficiency virus (HIV) antibody;
20. AAV neutralizing antibody titer >1:1000;
21. Those who are known to be allergic to the therapeutic drugs or diagnostic drugs used in the study protocol, including the investigational products, fluorescein sodium, indocyanine green, etc.;
22. Those who have used anticoagulant or antiplatelet drugs within 14 days before dosing;
23. Currently using or may need to use drugs that can cause crystal toxicity or retinal toxicity (such as deferrigin, chloroquine

    /hydroxychloroquine, tamoxifen, ethambutol, etc.);
24. Those who have a history of surgical operation within 1 month before screening, and/or currently have unhealed wounds (wound degree> stage III), moderate to severe ulcers, and fractures;
25. Patients with systemic infectious diseases requiring systemic treatment (oral, intramuscular or intravenous) at the time of screening;
26. Those who have received any AAV gene therapy products in the past;
27. Pregnant or lactating females;
28. Those who have participated in any clinical trial of drugs (excluding vitamins and minerals) within 3 months before screening;
29. Other those who need to be excluded in the opinion of the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs | 4 weeks
  Number and proportion of dose limited toxicity（DLTs）
Incidence of AEs | 52 weeks
  Number and severity of overall and ocular Adverse Events (AEs)
Incidence of SAEs | 52 weeks
  Number and severity of overall and ocular Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Visual function | 52 weeks
  Change from baseline in BCVA(Best Corrected Visual Acuity)(ETDRS)
OCT imaging | 52 weeks
  Change from baseline in CST(Central Retinal Thickness)(OCT)
the number of anti-VEGF remedy therapy | 52 weeks
  the number of anti-VEGF remedy therapy within 52 weeks after dosing;
mean annualized anti-VEGF injection rate | 52 weeks
  change in mean annualized anti-VEGF injection rate

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No